CLINICAL TRIAL: NCT06963593
Title: Efficacy and Safety of Nanosized Megestrol Acetate Combined With Immunochemotherapy in the Treatment of Anorexia and Cachexia in Advanced Gastric and Esophageal Cancer: A Randomized, Controlled, Multicenter Study
Brief Title: Clinical Study on the Treatment of Anorexia and Cachexia in Advanced Gastric and Esophageal Cancer With Nanosized Megestrol Acetate Combined With Immunochemotherapy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Chief Physician, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025YJZ29
Record Dates: First submitted 2025-04-10; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Advanced Gastroesophageal Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Megestrol Acetate Group (Experimental)
  Interventions: Drug: Nanocrystal Megestrol Acetate in Combination with First-Line Standard Immuno-Chemotherapy Regimen
- First-Line Standard Immuno-Chemotherapy Regimen (Other): Control Group
  Interventions: Drug: First-Line Standard Immuno-Chemotherapy Regimen

INTERVENTIONS:
Drug: Nanocrystal Megestrol Acetate in Combination with First-Line Standard Immuno-Chemotherapy Regimen — Megestrol Acetate Nanocrystal Oral Suspension Group: Nanocrystal Megestrol Acteate Oral Suspension (QD, up to 16 weeks from the initiation of immuno-chemotherapy) + PD-1 inhibitor (Q3W, until PD) + Chemotherapy regimen (TP regimen or XELOX regimen or SOX regimen selected based on cancer type, Q3W, as per package insert)
  Arms: Megestrol Acetate Group
Drug: First-Line Standard Immuno-Chemotherapy Regimen — PD-1 inhibitor (Q3W, until PD) + Chemotherapy regimen (TP regimen or XELOX regimen or SOX regimen selected based on cancer type, Q3W, as per package insert)
  Arms: First-Line Standard Immuno-Chemotherapy Regimen

SUMMARY:
This study is a prospective, randomized, parallel-controlled, multicenter clinical study. The purpose of this study is to evaluate the efficacy and safety of nanocrystalline megestrol acetate combined with the first-line standard immunochemotherapy regimen compared with the first-line standard immunochemotherapy regimen in the treatment of anorexia and cachexia in advanced gastric and esophageal cancer. Eligible patients with gastric and esophageal cancer will be randomly assigned in a 1:1 ratio to the nanocrystalline megestrol acetate combination group (referred to as the megestrol acetate group for short) or the first-line standard immunochemotherapy group (referred to as the standard control group for short).

ELIGIBILITY:
1. Aged between 18 and 75 years old, regardless of gender；
2. The Eastern Cooperative Oncology Group (ECOG) performance status score is 0-2；
3. The expected survival time is more than 3 months；
4. Good organ function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Quality of Life for Patients with Advanced Gastric Cancer and Esophageal Cancer | 1year
  Quality of Life Questionnaire (EORTC QLQ-C30; Physicians' Global Assessment score). The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30), a 30-item instrument, assesses health-related quality of life in cancer patients. The scale assesses 15 domains: 5 functional scales, 3 symptom scales, 6 single-item measures, and 1 global quality of life scale. Compared to baseline, a score change of ≥10 points in functional scales or the global quality of life scale indicates clinical significance (higher scores represent better functioning or quality of life). For symptom scales/single-item measures, a score increase ≥10 points signifies deterioration (higher scores indicate more severe symptoms or problems). An improvement is defined as either a ≥10-point increase in functional scale scores or a ≥10-point decrease in symptom scale scores.
Changes in Body Weight Relative to Baseline in Patients with Advanced Gastric and Esophageal Cancers | 1year
  1. Body weight (kg);
  2. Height (m);
  3. BMI (kg/m², calculated from weight and height).

SECONDARY OUTCOMES:
Impact on Survival Benefits in Patients with Advanced Gastric and Esophageal Cancers | 1year
  Progression-Free Survival
Impact on Survival Benefits in Patients with Advanced Gastric and Esophageal Cancers | 1year
  Overall Survival
Impact on Body Composition in Patients with Advanced Gastric and Esophageal Cancers | 1year
  L3-CT (Skeletal Muscle）
Impact on Body Composition in Patients with Advanced Gastric and Esophageal Cancers | 1year
  Appetite (Functional Assessment of Anorexia/Cachexia Therapy - Anorexia/Cachexia Subscale 12, FAACT-A/CS-12)